CLINICAL TRIAL: NCT05008276
Title: PANTHER Study: Puberty, Diabetes, and the Kidneys, When Eustress Becomes Distress
Brief Title: Puberty, Diabetes, and the Kidneys, When Eustress Becomes Distress (PANTHER Study)
Status: Recruiting | Type: Observational
Sponsor: Petter Bjornstad (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Seattle Children's Hospital (Other); University of Colorado, Denver (Other)
Responsible Party: Sponsor-Investigator, Petter Bjornstad, Assistant Professor, Seattle Children's Hospital
Organization: Seattle Children's Hospital (Other)
Other Study IDs: 21-3019
Record Dates: First submitted 2021-08-09; First posted 2021-08-17 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes Mellitus; Diabetic Kidney Disease; Adolescent Obesity; Pre Diabetes; Kidney Hypoxia; Puberty
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Nephropathies; Pediatric Obesity; Glucose Intolerance | interventions — p-Aminohippuric Acid; Iohexol; Dextrans

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — During the study, the investigators will collect blood and urine samples for assessment of kidney function and kidney injury markers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Youth with overweight/obesity and/or newly diagnosed T2D and elevated HbA1c: All participants will undergo GFR (Iohexol Inj 300 MG/ML), EPRF (Aminohippurate Sodium Inj 20%), Dextran sieving (Dextran 40 Sodium Inj 0.9%), IVGTT for insulin sensitivity, in addition to BOLD and ASL Kidney MRI
  Interventions: Drug: Aminohippurate Sodium Inj 20%; Drug: Iohexol Inj 300 MG/ML; Drug: Dextran 40
- Healthy normal-weight controls: All participants will undergo GFR (Iohexol Inj 300 MG/ML), EPRF (Aminohippurate Sodium Inj 20%), Dextran sieving (Dextran 40 Sodium Inj 0.9%), IVGTT for insulin sensitivity, in addition to BOLD and ASL Kidney MRI
  Interventions: Drug: Aminohippurate Sodium Inj 20%; Drug: Iohexol Inj 300 MG/ML; Drug: Dextran 40

INTERVENTIONS:
Drug: Aminohippurate Sodium Inj 20% — Diagnostic aid/agent used to measure effective renal plasma flow (ERPF)
  Other Names: Sodium 4-amino hippurate (PAH) inj 20% 2g/10mL; Para-aminohippurate; Aminohippuric acid
Drug: Iohexol Inj 300 MG/ML — Diagnostic aid/agent used to measure glomerular filtration rate (GFR)
  Other Names: omnipaque 300
Drug: Dextran 40 — Diagnostic aid/agent used to measure glomerular size and selectivity
  Other Names: Dextran Sieving

SUMMARY:
Early diabetic kidney disease (DKD) occurs in 50-70% of youth with type 2 diabetes (T2D) and confers high lifetime risk of dialysis and premature death. Youth-onset T2D typically manifests during or shortly after puberty in adolescents with obesity. Epidemiological data implicate puberty as an accelerator of kidney disease in youth with obesity and diabetes and the investigators posit that the link between puberty and T2D-onset may explain the high burden of DKD in youth-onset T2D. A better understanding of the impact of puberty on kidney health is needed to promote preservation of native kidney function, especially in youth with T2D.

DETAILED DESCRIPTION:
Puberty is a complex process of physiological changes, including neuroreproductive and growth hormone activation and rapid organ growth, that may predispose organs to injury. The kidneys may be especially susceptible because they are highly metabolically active and second only to the heart with respect to oxygen consumption per tissue mass. During puberty, the kidneys almost double in size, likely increasing the kidneys' already high energy expenditure. In parallel, puberty is associated with physiologic insulin resistance (IR), which is accentuated in obesity. Our central hypothesis is that obese youth with prediabetes and T2D experience relative kidney hypoxia during puberty due to a metabolic mismatch between increased energy expenditure and impaired substrate metabolism. In turn, the kidney hypoxia results in loss of glomerular charge and size selectivity leading to increased transglomerular transport of protein and kidney dysfunction. Our preliminary data showed that pubertal adolescents with obesity and/or diabetes exhibit relative kidney hypoxia compared to normal weight controls using functional magnetic resonance imaging (MRI) and that relative kidney hypoxia is greater in late vs. early puberty. However, determining the pubertal mechanisms contributing to kidney injury in youth with obesity and T2D requires serial evaluations throughout puberty. To assess the impact of pubertal changes within a 5-year study period, the investigators propose an accelerated longitudinal study design in which the investigators will enroll adolescents (8-14 years, 50% girls) with obesity and/or elevated hemoglobin A1c (HbA1c ≥6%) [n=60], and healthy normoglycemic controls [n=40] at Tanner (pubertal) stages 1-4 and examine them at baseline, 1 and 2-years. The investigators will then compare data by Tanner stage to construct an integrated portrayal of the physiological changes that occur throughout puberty. Given the rarity of T2D prior to pubertal onset, the investigators chose to enroll a high high-risk group: youth with obesity and/or HbA1c ≥6.0% to represent youth ranging from those at magnified risk of developing T2D to those recently diagnosed.

ELIGIBILITY:
Inclusion Criteria:

* HbA1c ≥6.0% for untreated high-risk group
* BMI ≥ 85th %ile for high-risk group
* Normal HbA1c ≤5.6% for control group
* Type 1 diabetes (T1D) Antibody negative

Exclusion Criteria:

* History of Chronic kidney disease (CKD) or acute kidney injury (AKI)
* Metabolic disorder prohibiting safe fasting
* Iodine or penicillin allergy
* Pregnancy
* Thrombophilia
* MRI contraindications
* Hormone therapy

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The investigators propose to address the specific aims of this study in an accelerated longitudinal project with 40 adolescents with normal HbA1c (≤5.6%) and 60 with overweight/obesity and/or newly diagnosed T2D (BMI≥85%ile) and elevated HbA1c (≥6.0%) or on anti-diabetic medications ranging from TS 1-4 (Ages 8-14 yr). They will be studied annually for 2 years.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-09-27 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Effective renal plasma flow (ERPF) | 3 Hours
  Measured by PAH Clearance
Glomerular Filtration Rate (GFR) | 3 hours
  Measured by iohexol clearance

SECONDARY OUTCOMES:
Insulin Sensitivity | 3 hours
  Measured by IV glucose tolerance test (IVGTT)
Renal perfusion | 10 min
  Arterial spin labeling (ASL) MRI
Renal oxygenation | 60 min
  Blood oxygen level dependent (BOLD) MRI

CONTACTS AND LOCATIONS:
Overall Officials: Petter Bjornstad, MD, Principal Investigator — University of Washington - Medicine Diabetes Institute
Locations (2):
- United States (2):
  - Children's Hospital Colorado, Aurora, Colorado
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided